CLINICAL TRIAL: NCT05373849
Title: Evaluation of the Efficacy of Aromatherapy on the Well-being of Hospital Healthcare Professionals: a Randomized Cross-over Trial
Brief Title: Evaluation of the Efficacy of Aromatherapy on the Well-being of Healthcare Professionals
Acronym: HERBAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier de la Region de Mulhouse et Sud Alsace (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: GHRMSA 1192; 2021-A02995-36 (Other: ANSM)
Record Dates: First submitted 2022-05-04; First posted 2022-05-13 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Healthcare Professionnals
Keywords: Aromatherapy; stress; anxiety; quality of life; critical care
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aromatherapy first then no intervention (Experimental): The participant will receive the study treatment (essential oils mixture in inhaler sticks for 2 months) and the control (no intervention for 2 months). At inclusion and at the end of each period, questionnaires of well-being, anxiety and stress will be completed
  Interventions: Dietary Supplement: essentiel oil mixtures in inhaler sticks (step 1) - no intervention (step 2); Dietary Supplement: no intervention (step 1) - essential oils mixture in inhaler sticks (step 2)
- No intervention first then Aromatherapy (Experimental): The participant will receive the control (no intervention for 2 months) and the study treatment (essential oils mixture in inhaler sticks for 2 months). At inclusion and at the end of each period, questionnaires of well-being, anxiety and stress will be completed.
  Interventions: Dietary Supplement: essentiel oil mixtures in inhaler sticks (step 1) - no intervention (step 2); Dietary Supplement: no intervention (step 1) - essential oils mixture in inhaler sticks (step 2)

INTERVENTIONS:
Dietary Supplement: essentiel oil mixtures in inhaler sticks (step 1) - no intervention (step 2) — The participant will receive the study treatment (essential oils mixture in inhaler sticks for 2 months) and the control (no intervention for 2 months). At inclusion and at the end of each period, questionnaires of well-being, anxiety and stress will be completed
Dietary Supplement: no intervention (step 1) - essential oils mixture in inhaler sticks (step 2) — The participant will receive the control (no intervention for 2 months) and the study treatment (essential oils mixture in inhaler sticks for 2 months). At inclusion and at the end of each period, questionnaires of well-being, anxiety and stress will be completed.

SUMMARY:
The main objective is to evaluate the efficacy of aromatherapy (inhaler sticks) on the well-being of healthcare professionals practicing in medical and surgical intensive care unit, operating room/anesthesia and emergency departments

DETAILED DESCRIPTION:
The secondary objectives of this study are :

1. To evaluate the efficacy of aromatherapy on anxiety of healthcare professionals;
2. To evaluate the efficacy of aromatherapy on stress symptoms of healthcate professionals;
3. To assess compliance with aromatherapy.

Conduct of research:

All participants included in the study will receive the study treatment (essential oils mixtures in inhaler sticks for 2 months) and the control (no intervention for 2 months), in random order. At inclusion and at the end of each period, questionnaires of well-being, anxiety and stress will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare professional ;
* Working in a medical or surgical intensive care unit or in a operating room/anesthesia unit or in the emergency department;
* Agrees not to use any topical, oral or inhaled essential oils during the two study periods, other than those specified in the study protocol;
* Written informed consent;

Exclusion Criteria:

* Pregnant or breastfeeding woman;
* Known allergies to essential oils;
* Asthma;
* Scheduled departure from the unit;
* Antidepressant treatment or anxiolytic treatment;
* Taking topical, oral or inhaled essential oils durink the week prior to inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
World Health Organization index of well-being | Through study completion, 4 months
  The World Health Organization well-being index consists of 5 items with 6 response modalities distributed on a frequency scale from 0 to 5. A global score is obtained by adding the answers to the 5 items, then multiplying this result by 4, i.e. a global score varying from 0 to 100. 0 is the worst score possible and 100 is the best score possible.

SECONDARY OUTCOMES:
Spielberger General Anxiety Questionnaire | Through study completion, 4 months
  The Spielberger General Anxiety Questionnaire consists of 20 items with 4 response modalities distributed on a frequency scale from 1 to 4 (the scoring of some questions being reversed). A global score between 20 and 80 is obtained by adding the answers to the 20 items.
  For women the average score is 47.13.For men the average score is 39.27. A score above these averages indicates an anxious personality. The higher the score, the greater the anxiety. For men, a score higher than 51 indicates significant anxiety that interferes with quality of life. For women, a score higher than 61 indicates significant anxiety that interferes with quality of life.
Perceived Stress Scale | Through study completion, 4 months
  The Perceived Stress Scale is a 10-item scale with 5 response modalities distributed on a frequency scale from 0 to 4 (the scoring of some questions being reversed). A global score between 0 and 40 is obtained by adding the answers to the 10 items.
  Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress
Follow-up diary | End of aromatherapy, 2 months
  Compliance collected using a follow-up diary in which the participant will enter the average daily use of the "rest" stick and the "work" stick over the past week

CONTACTS AND LOCATIONS:
Locations (1):
- GHRMSA, Mulhouse, France

REFERENCES:
- [Derived] Anne-Florence D, Samuel D, Cindy P, Marie D, Clement P. The Efficacy of Aromatherapy on Well-Being and Stress. Nurs Crit Care. 2026 Jan;31(1):e70270. doi: 10.1111/nicc.70270. PMID 41330862